CLINICAL TRIAL: NCT03978286
Title: Vortioxetine Versus Sertraline in Control Metabolic, Distress and Depression in Mexican Patients With Type 2 Diabetes
Brief Title: Vortioxetine vs Sertraline in Mexicans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Juárez Autónoma de Tabasco (Other)
Responsible Party: Principal Investigator, ISELA ESTHER JUAREZ-ROJOP Ph.D., Principal Investigator, Universidad Juárez Autónoma de Tabasco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00228/16.
Record Dates: First submitted 2019-03-18; First posted 2019-06-07 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Depression; Type 2 Diabetes Mellitus
Keywords: depression; Type 2 diabetes Mellitus; vortioxetine; sertraline
MeSH Terms: conditions — Depression; Diabetes Mellitus, Type 2 | interventions — Vortioxetine; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vortioxetine therapy (Experimental): patients who gave informed consent and met the inclusion criteria were attended by a psychiatrist. The pharmacological management were randomly assigned: these group of patients received vortioxetine (10 mg/day) for 8 weeks, in addition, the patients maintained their anti-diabetic treatment (oral hypoglycemic or insulin)
  Interventions: Drug: Vortioxetine
- Sertraline therapy (Experimental): patients who gave informed consent and met the inclusion criteria were attended by a psychiatrist. The pharmacological management were randomly assigned: these group of patients received sertraline (75 mg / day) for 8 weeks, in addition, the patients maintained their anti-diabetic treatment (oral hypoglycemic or insulin)
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Vortioxetine — 10 mg per day
  Other Names: Brintellix
  Arms: Vortioxetine therapy
Drug: Sertraline — 75 mg per day
  Other Names: zoloft
  Arms: Sertraline therapy

SUMMARY:
Depression in patients with type 2 diabetes is often undiagnosed and remains untreated, leading to poor therapy adherence and ill health-related outcomes. The aim of study was evaluated the effect of vortioxetine versus sertraline in the treatment of depression, diabetes-related distress and control metabolic in subjects with type 2 diabetes and depression. was included patients who were glycosylated hemoglobin ≥ 7.5%, 18 to 60 years of age and written consent . Pharmacological treatment for depression was assigned randomly: vortioxetine (10 mg/day) or sertraline (75 mg/day) for 8 weeks. Biochemical parameters, anthropometric measures and depression symptoms were evaluated before and at the and at the 8 weeks after antidepressant treatment.

DETAILED DESCRIPTION:
The assessment consisted of an extended face-to-face interview. The patients answered a structured questionnaire used to collect: sociodemographic characteristics (gender, age, education, occupation and marital status) and clinical data (pharmacotherapy, habits, consumed of drugs, diabetes complications and comorbidities). Depression was screened using Hamilton Depression Rating Scale score ≥ 14 (HAM-D), Center for epidemiologic studies depression scale revised in Spanish (CES-DR35), and Problem Areas in Diabetes Questionnaire (PAID-V); anthropometrics measurements were evaluated (weight, waist circumference and body mass index). Besides, blood samples were drawn for the following biochemical parameters: fasting plasma glucose, glycated hemoglobin (HbA1c), cholesterol and triglycerides. Patients who gave informed consent and convened inclusion criteria were attended by a psychiatrist. The pharmacological management were randomly assigned: vortioxetine (10 mg/day) or sertraline (75 mg/day) for 8 weeks, in addition, the patients maintained their established anti-diabetic treatment (oral hypoglycemic or insulin). The study ended at the 8th week, subjects were attended by psychiatrist and blood samples were drawn for evaluated biochemical parameters and the structured questionnaire previously described was applicated.The clinical measures and biochemical parameters were done baseline and after 8-week pharmacological treatment. Finally the effect of both antidepressants were compared.

ELIGIBILITY:
Inclusion Criteria:

* Individuals had to be between 18 and 85 years of age
* Clinical diagnosis of type 2 diabetes mellitus based on the American Diabetes Association criteria,
* They had to receive anti-diabetic treatment, Clinical diagnosis of major depressive episode according Association Diagnostic and Statistical Manual of Mental Disorders, five edition (DSM-V)
* Ratings scale score ≥ 14 by means of Hamilton Depression scale (HAM-D)
* Patients had to give verbal and written informed consent for this study

Exclusion Criteria:

* Neurological illness
* Psychoactive medications
* Type I diabetes
* Active suicidal ideation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Effect of antidepressant treatment (sertraline versus vortioxetine) in remission of depression in depressed type 2 diabetic patients. | 8 weeks
  Two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The assessment of depression was performed by the Hamilton Depression Rating Scale (HAM-D) validated in the Spanish version. We used a 17-item reduced version, the range of scale was 0-50, includes the following items: psychic anxiety, somatic anxiety, gastrointestinal somatic symptoms, general somatic symptoms, hypochondriasis, and insight. A score of 8 and above indicates depression and a high levels of anxiety symptoms. Where 14 was the cutoff point of this scale; patients with this score were diagnosed with major depression and included in the study. Depression was screened using HAM-D at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.
Effect of antidepressant treatment (sertraline versus vortioxetine) in severity of depression in depressed type 2 diabetic patients. | 8 weeks
  Two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The severity of depression was measured with the center for epidemiologic studies depression scale revised in Spanish (CES-DR35). Previous studies in a Mexican population reported a Cronbach α score of 0.9. This questionnaire consists of 35 items, the range of scale was 0-140, among them are: depressed mood, anhedonia, appetite, sleep problem, psychomotor retardation, fatigue, guilt/conscience, thinking, suicidal ideation and social. A score of 16 and above indicates clinically significant symptoms of major depression episode and the severity of depression. Depression was screened using CES-DR35 at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.
Effect of antidepressant treatment (sertraline versus vortioxetine) in treatment of diabetes related stress in depressed type 2 diabetic patients. | 8 weeks
  Two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. Diabetes related stress was screened using 5-item Problem Areas in Diabetes Scale (PAID-5). The scale gives a total score from 0 to 20. A score of 8 and above indicates a high level of diabetes-related distress. Diabetes related stress was screened using PAID-5 at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.
Effect of antidepressant treatment (sertraline versus vortioxetine) in fasting plasma glucose level in depressed type 2 diabetic patients. | 8 weeks
  Two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The glycemic variable was measured by fasting plasma glucose level in mg/dl. at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.
Effect of antidepressant treatment (sertraline versus vortioxetine) in glycemic control in depressed type 2 diabetic patients. | 8 weeks
  Two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The glycemic variable was measured by glycosylated hemoglobin A 1c in percentage at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.
Effect of antidepressant treatment (sertraline versus vortioxetine) in cholesterol control in depressed type 2 diabetic patients. | 8 weeks
  Two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The metabolic variable was measured by cholesterol in mg/dL at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.
Effect of antidepressant treatment (sertraline versus vortioxetine) in triglycerides control in depressed type 2 diabetic patients. | 8 weeks
  Two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The metabolic variable was measured by triglycerides in mg/dL at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.

SECONDARY OUTCOMES:
Effect of antidepressant treatment (sertraline versus vortioxetine) in weigh in depressed type 2 diabetic patients. | 8 weeks
  two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The anthropometric variables were evaluated in the weight in kilograms at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.
Effect of antidepressant treatment (sertraline versus vortioxetine) in waist circumference in depressed type 2 diabetic patients. | 8 weeks
  two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The anthropometric variables were evaluated in waist circumference in centimeters at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.
Effect of antidepressant treatment (sertraline versus vortioxetine) in anthropometric variables in depressed type 2 diabetic patients. | 8 weeks
  two groups of depressed type 2 diabetic patients were involve in the study: one group received sertraline and the second vortioxetine. The anthropometric variables were evaluated, weight and height will be combined to report BMI in kg/m^2 at the beginning of the study and at 8 weeks of treatment. Finally the effect of both antidepressant were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Isela Juarez Rojop, Ph.D, Principal Investigator — Universidad Juárez Autonoma de Tabasco

IPD SHARING:
Plan to Share IPD: Yes
the information will be available when contacting the correspondence author
Supporting Information: SAP, ICF, CSR
Time Frame: Once the article is published, information about the study will be available for a period of 3 years.
Access Criteria: direct contact with the correspondence author

REFERENCES:
- [Background] Petrak F, Herpertz S, Albus C, Hermanns N, Hiemke C, Hiller W, Kronfeld K, Kruse J, Kulzer B, Ruckes C, Zahn D, Muller MJ. Cognitive Behavioral Therapy Versus Sertraline in Patients With Depression and Poorly Controlled Diabetes: The Diabetes and Depression (DAD) Study: A Randomized Controlled Multicenter Trial. Diabetes Care. 2015 May;38(5):767-75. doi: 10.2337/dc14-1599. Epub 2015 Feb 17. PMID 25690005
- [Background] Rachdi C, Damak R, Fekih Romdhane F, Ouertani H, Cheour M. Impact of sertraline on weight, waist circumference and glycemic control: A prospective clinical trial on depressive diabetic type 2 patients. Prim Care Diabetes. 2019 Feb;13(1):57-62. doi: 10.1016/j.pcd.2018.09.003. Epub 2018 Oct 2. PMID 30287230
- [Background] D'Agostino A, English CD, Rey JA. Vortioxetine (brintellix): a new serotonergic antidepressant. P T. 2015 Jan;40(1):36-40. PMID 25628505
- [Background] Chokka P, Bougie J, Rampakakis E, Proulx J. Assessment in Work Productivity and the Relationship with Cognitive Symptoms (AtWoRC): primary analysis from a Canadian open-label study of vortioxetine in patients with major depressive disorder (MDD). CNS Spectr. 2019 Jun;24(3):338-347. doi: 10.1017/S1092852918000913. Epub 2018 May 24. PMID 29792585
- [Background] Kesim M, Tiryaki A, Kadioglu M, Muci E, Kalyoncu NI, Yaris E. The effects of sertraline on blood lipids, glucose, insulin and HBA1C levels: A prospective clinical trial on depressive patients. J Res Med Sci. 2011 Dec;16(12):1525-31. PMID 22973359
- [Background] Llorca PM, Lancon C, Brignone M, Rive B, Salah S, Ereshefsky L, Francois C. Relative efficacy and tolerability of vortioxetine versus selected antidepressants by indirect comparisons of similar clinical studies. Curr Med Res Opin. 2014 Dec;30(12):2589-606. doi: 10.1185/03007995.2014.969566. Epub 2014 Oct 10. PMID 25249164
- [Background] Petrak F, Baumeister H, Skinner TC, Brown A, Holt RIG. Depression and diabetes: treatment and health-care delivery. Lancet Diabetes Endocrinol. 2015 Jun;3(6):472-485. doi: 10.1016/S2213-8587(15)00045-5. Epub 2015 May 17. PMID 25995125
- [Background] Rosenblat JD, Kakar R, McIntyre RS. The Cognitive Effects of Antidepressants in Major Depressive Disorder: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Int J Neuropsychopharmacol. 2015 Jul 25;19(2):pyv082. doi: 10.1093/ijnp/pyv082. PMID 26209859
- [Derived] Tovilla-Zarate CA, Perez-Mandujano A, Ramirez-Gonzalez IR, Fresan A, Suarez-Mendez S, Martinez-Villasenor E, Rodriguez-Sanchez E, Villar-Soto M, Lopez-Narvaez ML, Gonzalez-Castro TB, Ble-Castillo JL, Juarez-Rojop IE. Vortioxetine versus sertraline in metabolic control, distress and depression in Mexican patients with type 2 diabetes. Ann Transl Med. 2019 Nov;7(22):656. doi: 10.21037/atm.2019.10.56. PMID 31930057